CLINICAL TRIAL: NCT02683343
Title: The Use of Ultrasound to Quantify Muscle Overlying the Carpal Tunnel
Status: Withdrawn | Type: Observational
Why Stopped: PI is away, will hopefully perform the study at another institution.
Sponsor: Clalit Health Services (Other)
Responsible Party: Sponsor
Other Study IDs: Muscle mass
Record Dates: First submitted 2015-08-16; First posted 2016-02-17 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2015-07

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- carpal tunnel syndrome: No intervention
- normals: no intervention

SUMMARY:
Carpal tunnel syndrome (CTS) is a common condition that still lacks a reliable, objective screening test. Many anatomical aspects of the syndrome have been studied including the dimensions of the carpal tunnel and shape of the nerve within the tunnel. The investigators have observed varying amounts of muscle overlying the carpal tunnel in patients undergoing surgery for the condition. Assuming that this muscle may have a dynamic role in the development of the condition, the investigators attempted to quantify this muscle using ultrasound (US).

The purpose of this study was to devise a technique to evaluate the amount of muscle overlying the carpal tunnel.

The hypothesis is that patients with carpal tunnel syndrome will have significantly more muscle overlying the carpal tunnel than individuals without carpal tunnel syndrome.

DETAILED DESCRIPTION:
Introduction:

The pathophysiology of carpal tunnel syndrome (CTS) is in all probability multifactorial including many parameters that ultimately increase the pressure within the carpal tunnel. It is likely that the increased pressure then causes injury to the median nerve and the signs and symptoms of CTS. The relationship between the size or dimensions of the hand and the occurrence of CTS has been evaluated and "square-shaped" hands have also been examined to determine if there is an increased tendency to develop CTS. The literature remains inconclusive at this time. Other static anatomical parameters that have been evaluated include the size of the carpal tunnel and the thickness and biomechanical properties of the transverse carpal ligament again without absolute consensus in the literature.

Additional studies have evaluated the role of the intrinsic musculature within and surrounding the carpal tunnel in the etiology of CTS. Most of these studies have evaluated the muscles as space occupying lesions that add to the pressure within the carpal tunnel. The investigators believe that some of the muscles described, specifically those that are found within the transverse carpal ligament and that cross the area of the carpal tunnel, actually have a dynamic role in the etiology of CTS, especially in manual laborers that use their hands in a forceful manner in a repetitive fashion. It is also possible that this anatomic variant (muscles crossing the area of the carpal tunnel) is related to the "square "hand configuration and that this dynamic contribution to the pressure within the carpal tunnel is the reason for the increased incidence of CTS in these patients. The purpose of this study is to quantify the amount of muscle crossing the area of the carpal tunnel in normal individuals and to compare it to the amount of muscle in the wrists of patients with CTS.

Hypothesis: Participants with CTS will have more muscle crossing the carpal tunnel that normal controls (without CTS).

Purpose: To compare the amount of muscle crossing the carpal tunnel in normal controls (without CTS) and in patients with CTS

Specific aims:

1. To develop a system to quantify the amount of muscle crossing the carpal tunnel area using ultrasound of the wrist area.
2. To compare this measurement in normal wrists and in wrists with CTS
3. To compare the measurements in the CTS patients to intraoperative evaluation of the amount of muscle crossing the carpal tunnel area .
4. To compare these measurements to the external measurements of the hand (palm width/palm length)

Methods:

Fifty participants will be recruited for the study. Twenty five participants with no CTS- and twenty five with CTS.

The CTS group inclusion criteria:

The diagnosis of CTS will include:

1. Signs and symptoms of CTS: nighttime numbness and tingling or numbness and tingling in a median nerve distribution with a positive phalen or tinel or forearm compression test
2. A nerve conduction test and electromyography (NCT and EMG) that is positive for CTS.

The participants without CTS inclusion criteria:

1) Individuals that do not have any signs and or symptoms of CTS.

Exclusion criteria:

1. Individuals that have a known history of peripheral neuropathy or other condition in the hand including recent significant trauma.
2. Patients with incomplete or unclear evaluation and tests.
3. Individuals unwilling to sign a consent form to participate in the study.

Patients that meet the inclusion criteria and that are sent for carpal tunnel release surgery will be consented and examined on the day of surgery. Their US results, external palmar measurements as well as the amount of overlying muscle will be recorded as well as demographic data. Demographic information, occupational history, history of hand diagnoses and procedures as well as history pertinent to CTS (nighttime numbness and tingling, pain, perceived pinch weakness, and duration of symptoms) will be collected. Results of nerve conduction testing (NCT) will be recorded.

Physical examination findings pertinent to CTS will be collected including pinch strength, grip strength, 2-point discrimination, and the hand measurements of palm width (PW), palm length (PL).

External measurements: PL is measured as the vertical length from the midline of the distal wrist crease to the proximal middle finger. PW is measured as the horizontal length from the base of the 1st metacarpophalangeal (MP) joint along the proximal palmar crease.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of CTS will include signs and symptoms of CTS: nighttime numbness and tingling or numbness and tingling in a median nerve distribution with a positive phalen or tinel or forearm compression test as well as a nerve conduction test and electromyography (NCT and EMG) that is positive for CTS.
* The normal subjects: individuals that do not have any signs and or symptoms of CTS.

Exclusion Criteria:

* Patients or individuals that have a known history of peripheral neuropathy or other condition in the hand including recent significant trauma.
* Patients with incomplete or unclear evaluation and tests.
* Individuals unwilling to sign a consent form to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with the diagnosis of CTS and those without
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
amount-depth of muscle overlying the carpal tunnel | 2 years
  As determined by ultrasound